CLINICAL TRIAL: NCT05489406
Title: Relative Bioavailability Study to Investigate a Potential Interaction Between Dolutegravir (DTG) and Tenofovir Alafenamide Fumarate/Emtricitabine (F/TAF) Administered as Paediatric Tablet Formulations
Brief Title: Relative Bioavailability Study to Investigate a Potential Interaction Between DTG DT and F/TAF TOS.
Acronym: UNIVERSALRBA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UNIVERSAL RBA
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single-dose DTG 30 mg (Active Comparator): Healthy volunteers receiving a single-dose DTG 30 mg as 6X5 mg dispersible tablets (DT) as a dispersed suspension in a fasted state. Samples will be taken pre-dose (t=0) and 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, and 48 hours post ingestion.
  Interventions: Drug: DTG DT (6 x 5 mg)
- Single-dose F/TAF 180/22.5 mg (Active Comparator): Healthy volunteers receiving a single-dose F/TAF 180/22.5 mg as 3X60/7.5 mg TOS as a dispersed suspension in a fasted state. Samples will be taken pre-dose (t=0) and 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, and 48 hours post ingestion.
  Interventions: Drug: F/TAF TOS (3 x 60/7.5 mg)
- Single-dose DTG 30 mg and F/TAF 180/22.5 mg (Experimental): Healthy volunteers receiving a single-dose F/TAF 180/22.5 mg as 3X60/7.5 mg TOS + DTG 30 mg as 6X5 mg DT as a co-dispersed suspension in a fasted state. Samples will be taken pre-dose (t=0) and 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, and 48 hours post ingestion.
  Interventions: Drug: DTG DT (6 x 5 mg); Drug: F/TAF TOS (3 x 60/7.5 mg)

INTERVENTIONS:
Drug: DTG DT (6 x 5 mg) — DTG 5mg dispersible tablet
  Other Names: Tivicay 5 mg (ViiV)
  Arms: Single-dose DTG 30 mg; Single-dose DTG 30 mg and F/TAF 180/22.5 mg
Drug: F/TAF TOS (3 x 60/7.5 mg) — 60/7.5 mg TOS emtricitabine/TAF
  Other Names: F/TAF TOS 60/7.5 mg (Gilead)
  Arms: Single-dose DTG 30 mg and F/TAF 180/22.5 mg; Single-dose F/TAF 180/22.5 mg

SUMMARY:
This relative bioavailability (RBA) study will be conducted to investigate whether there is a potential pharmacokinetic effect when paediatric DTG and F/TAF are taken together as dispersible formulations. This study will be performed in healthy volunteers instead of HIV-infected patients.

DETAILED DESCRIPTION:
This relative bioavailability (RBA) study will be conducted to investigate whether there is a potential pharmacokinetic effect when paediatric DT DTG (30 mg dose) and F/TAF TOS (180/22.5 mg dose) are taken together. For this purpose, Gilead's F/TAF 60/7.5 mg TOS tablets and ViiV Healthcare's DTG 5 mg tablets will be used. Given the very low plasma concentration of TAF (very probably mainly under the detection limit) with a single dose of 7.5 mg in adults, 3 tablets of F/TAF 60/7.5 mg (180/22.5 mg) will be given, which is similar to the adult dose. It was considered to keep the ratio between DTG and F/TAF similar to the to be developed paediatric fixed dose combination tablet, which would have resulted in a DTG dose of 60mg DTG DT. But because DTG shows nonlinear kinetics above a dose of 50 mg FCT (3), it was decided to use DTG 30 mg DT tablets, which is bioequivalent to adult dose of 50 mg FCT. For all compounds, a dose similar to the adult dose will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 and not older than 55 years of age at the day of screening.
2. Subject weighs at least 40 kg.
3. Subject has a BMI of 18.5-30 kg/m2, extremes included.
4. Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
5. Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, haematology and urinalysis testing within four weeks prior to day 1. Results of biochemistry, haematology and urinalysis testing should be within the laboratory's reference ranges. If laboratory results are not within the reference ranges, the subject is included based on the Investigator's judgment that the observed deviations are not clinically relevant. This should be clearly recorded.
6. Subject has a normal blood pressure and pulse rate, according to the Investigator's judgment.
7. Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to day 1.

Exclusion Criteria:

1. Positive HIV test.
2. Positive hepatitis B or C test.
3. Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
4. Relevant history or current condition that might interfere with drug absorption, distribution, metabolism, or excretion.
5. Inability to understand the nature and extent of the study and the procedures required.
6. Pregnant female (as confirmed by an hCG test performed less than 4 weeks before day 1) or breast-feeding female. Female subjects of childbearing potential without adequate contraception, e.g., hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the study.
7. Therapy with any drug (including herbal remedies, multivitamins, iron supplements and calcium supplements) for two weeks preceding day 1, except for acetaminophen.
8. Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal disorders (renal failure determined as an estimated Glomerular Filtration Rate (eGFR) below 50 ml/min (MDRD-based)), hepatic disorders (Child-Pugh B or C), hormonal disorders (especially diabetes mellitus), coagulation disorders.
9. History of or current abuse of drugs, alcohol or solvents.
10. Participation in a drug study within 60 days prior to day 1. 11. Donation of blood within 60 days prior to day 1.

12. Febrile illness within 3 days before day 1. 13. Co-worker of Radboud university medical center.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
The relative bioavailability of TAF and TFV | 17 days
  The relative bioavailability of TAF and TFV after a single-dose F/TAF 180/22.5 mg as 3X60/7.5 mg TOS (reference TAF) compared to TAF and TFV after a single-dose F/TAF 180/22.5 mg as 3X60/7.5 mg TOS in combination with a single dose of DTG 30 mg as 6X5 mg DT tablets (test).
The relative bioavailability of FTC | 17 days
  The relative bioavailability of FTC after a single-dose F/TAF 180/22.5 mg as 3X60/7.5 mg TOS (reference FTC) compared to FTC after a single-dose F/TAF 180/22.5 mg as 3X60/7.5 mg TOS in combination with a single dose of DTG 30 mg as 6X5 mg DT tablets (test).
The relative bioavailability of DTG | 17 days
  The relative bioavailability of DTG after a single-dose DTG 30 mg as 6X 5 mg DT tablets (reference DTG) compared to DTG after a single-dose F/TAF 180/22.5 mg as 3X60/7.5 mg TOS in combination with a single dose of DTG 30 mg as 6X5 mg DT tablets (test).
The relative bioavailability of the potential interaction and pharmacokinetics | 17 days
  The relative bioavailability of the potential interaction, the pharmacokinetics (AUC0-∞, Cmax, Tmax, T1⁄2) of DTG, FTC, TAF and TFV will be obtained and the geometric mean ratios of the AUC0-tlast (TAF), AUC0-∞ (DTG, FTC and TFV only), Cmax , and Cmin (DTG, FTC and TFV only) of the test versus reference treatment

SECONDARY OUTCOMES:
Adverse events | 17 days
  Adverse events will be described and compared (including clinically relevant laboratory abnormalities) of the treatments with F/TAF and DTG once daily.

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, Prof.dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- RTCCS Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No